CLINICAL TRIAL: NCT03563456
Title: Development of Structured Exercise Program Based on Patient Condition for Type 2 Diabetes Mellitus Management
Brief Title: Development of Structured Exercise Program for T2DM Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Nani Cahyani Sudarsono, Vice Head of Center for Sports and Exercise Studies, Indonesian Medical Education and Research Center, Faculty of Medicine, Universitas Indonesia (Indonesia University), Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FKUI 17-05-0554
Record Dates: First submitted 2018-05-24; First posted 2018-06-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Type 2 Diabetes Mellitus; High-Intensity Interval Training; Resistance Training; Oxidative Stress; Physical Fitness
Keywords: structured exercise; glycemic control; Type 2 Diabetes Mellitus; interval training; resistance training; oxydative stress; physical fitness
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The assessors for blood measure are not aware of the group of experiment, since the blood samples will not carry any descriptions of the group.
  The assessors for physical fitness are not aware of the group of experiment, since the medical record is not provided to the assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERIMENT (EXP) (Experimental): Subjects conduct the structured combined exercise in form of combination of High Intensity Interval Training and Resistance Training
  Interventions: Behavioral: structured combined exercise
- CONTROL (KTR) (Active Comparator): Subjects conduct structured exercise of cardiorespiratory training in form of lower-volume continuous cardiorespiratory exercise.
  Interventions: Behavioral: cardiorespiratory exercise

INTERVENTIONS:
Behavioral: structured combined exercise — A structured designed exercise consists of three times per week interval cardiorespiratory training of High Intensity Interval Training incorporates cycles of 1:4 interval and two times per week Resistance Exercise consists of nine-movement.
  Arms: EXPERIMENT (EXP)
Behavioral: cardiorespiratory exercise — Once per week continuous cardiorespiratory training of moderate intensity
  Arms: CONTROL (KTR)

SUMMARY:
The study started by the process of designing a structured exercise that will manage the T2DM with regards to the effectiveness in glycemic control, the benefit for physical fitness, and safe. Subjects consist of 18 - 65 years old T2DM patients are allocated into 2 groups; EXP group and KTR group. The EXP group follow the protocol of 12-week structured exercise, combination of 3 times per week high intensity interval training with 2 times per week resistance exercises. The pre- and post- measure are physical fitness consists of VO2max, grip strength, sit and reach, push ups, back extension, BMI and body fat percentage; HbA1c; plasma MDA and SOD. The KTR group follow the once a week continuous exercise program. The structured exercise is hypothesized to lower HbA1c, lower plasma MDA, increase SOD.

DETAILED DESCRIPTION:
A structured exercise program is developed incorporating cardiorespiratory and resistance exercise. The cardio-respiratory exercise is interval training (High Intensity Interval Training/HIIT), combination of one-minute High Intensity Exercise (HIE) and four-minute Low Intensity Exercise aiming for six cycles per exercise session at the end of the program. The resistance exercise consist of nine exercises, covers knee extension (leg raise), shoulder press, chair squat, back row, chest press, lateral pull down, hamstring curl, back up, and crunches. The program is to enable subjects to do all the exercises without any major complains, therefore the load is increased gradually. At start, the first two weeks consists of 20-minute continuous cardiorespiratory exercise at 60-70% HR max on treadmill and nine resistance exercise using no weight or minimal external weight. From the third week, the interval training will begin with four cycles of one-minute HIE at 90% HRmax followed by four-minute LIE at 70% HRmax. The resistance exercises are then beginning with one set of light eight-repetition for each exercise. The training load of interval training will increase at the seventh week to reach the target of HIE at 92% HRmax followed by four-minute LIE at 75% HRmax. The resistance exercises progress with one set of 10-repetition of light resistance at week 3-6, then two sets of 10-repetition of medium to heavy resistance.

The subjects are recruited from the diabetes registry at primary care clinics near the exercise facility. The patients are contacted and going through screening examinations such as physical examination including Blood Pressure and ECG recording; fundus photography; blood examination for HbA1c, Hb, and and urine examination for albumin and creatinine measurement.

The eligible subjects will the follow the initial examination to determine the level of physical fitness (cardiorespiratory fitness, muscle strength, muscle endurance, flexibility, and body composition measures); plasma MDA and SOD; HbA1c; and Quality of Life (QoL) measure.

Two groups will be formed, the experiment (EXP), and control (KTR) groups using block of four random allocation. Twelve-week structured exercise program is conducted under physician supervision. For each exercise session, the eligibility criteria is resting HR not more than 100/min; resting BP not more than 180/100 mmHg, and glucose level not more than 300 mg/dL. The subjects are also advised to report any adverse feelings or if they perceived untolerable exertion.

The EXP group program consists of three-session per week of cardiorespiratory interval training and two-session per week of resistance exercise. The KTR group program consists of once per week of continuous cardiorespiratory exercise. The program for the KTR group is also a progression of duration and intensity from 20-minute 60-70% HRmax to 30-minute 75-80% HRmax at the last six week of the program.

During the 12-week program, the subjects are asked to maintain their medication, diet, and physical activities. All of the subjects carry a pedometer during the 12-week program, and the diet and physical activities are to be recorded at the end of each 4-week time using three-day food record and Bouchard's three-day physical activity record.

At the end of the program, the examination to determine the level of physical fitness (cardiorespiratory fitness, muscle strength, muscle endurance, flexibility, and body composition measures); plasma MDA and SOD; HbA1c; and Quality of Life (QoL) measure are repeated. The EXP-KTR group mean difference and the difference of increase/decrease between group are measured to determine the effect of the program.

To ensure about the effect of the program, the influence of nutrition intake and physical activity to the primary results will be analyzed. So as the influence of other independent factors such as gender, age, and the previous history of length of diagnosed as T2DM and regular physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Registered as type 2 Diabetes Mellitus for more than 6 months in primary care clinics
* Medication: oral anti hyperglycemic agent
* Glucose controlled shows by HbA1c not more than 10.5%
* Able to move around without assisstant
* Commit to do three times per week of exercise at the training center for 12-week
* Voluntarily sign an informed consent document

Exclusion Criteria:

* Already developing type 2 Diabetes Mellitus complications, such as severe microalbuminuria, severe non proliferative diabetes retinopathy
* Have medical condition that prevent oneself from doing exercise, such as history of chest pain/miocardial infarction, exercise-induced asthma, scoliosis, severe arthritis

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Glycemic control (HbA1c) | Change from baseline HbA1c (%) after 12 weeks of exercise
  The percentage of glycated hemoglobin
Maximum oxygen uptake (VO2max) | Change from baseline VO2max (ml/kg.min) after 12 weeks of exercise
  Maximum volume of oxygen uptake per kilogram of body weight per minute (ml/kg.min) as part of physical fitness measure.
Grip strength | Change from baseline Grip strength (kg) after 12 weeks of exercise
  A measure of isometric hand strength shown by maximum force applied by the hand to squeeze a part of grip dynamometer (kilogram) as part of physical fitness measure.
Push-up | Change from baseline Push-up (number) after 12 weeks of exercise
  A measure of muscular endurance of the chest, shoulders and arms, shown by the number of as many consecutive push-ups performed without time limit as part of physical fitness measure.
Sit and reach | Change from baseline Sit and reach (cm) after 12 weeks of exercise
  A measure of general flexibility shown by hamstring and lower back flexibility, as a result of maximum flexion of the upper body with legs fully extended, arms evenly stretched with palms down and hands together reaching forward as far as possible (centimeter) as part of physical fitness measure.
Back extension | Change from baseline Back extension (sec) after 12 weeks of exercise
  A measure of the isometric endurance (time in seconds) of the trunk extensor muscles, as a result of maintaining horizontal position while lie face down (seconds) as part of physical fitness measure.
BMI (Body Mass Index) | Change from baseline BMI (kg/m^2) after 12 weeks of exercise
  A measure of body composition based on weight (kilogram) in relation to height (meter), combined to report in kg/m^2 as part of physical fitness measure
Fat percentage | Change from baseline Fat percentage (kg/m^2) after 12 weeks of exercise
  A measure of fat percentage using bio-electrical impedance analysis to measure body fat (percent) as part of physical fitness measure.
Free radicals | Change from baseline MDA (nmol/mL) after 12 weeks of exercise
  The measure of production of the free radicals, as a result of measuring concentration (nmol/mL) of plasma malondialdehyde (MDA) as part of oxydative stress measure.
Antioxydants | Change from baseline SOD (U/mL) after 12 weeks of exercise
  The measure of antioxydants activities, as a result of measuring plasma superoxide dismutase (SOD) activity (U/mL) as part of oxydative stress measure.

SECONDARY OUTCOMES:
Quality of Life | Before and after 12-week intervention
  A measure of health-related quality of life using visual analog scale (VAS) part of EuroQol Group EQ-5D questionnaire, ranging of scale 0 - 100 (0 is the worst health state and 100 is the best health state that the subject can imagine)
Physical activity during intervention | 4th, 8th, and 12th week of intervention
  The amount of energy expenditure during intervention, conducted by records of steps stated by each subject's pedometer and in accordance with Bouchard's three-day physical activity record
Nutritional intake during intervention | 4th, 8th, and 12th week of intervention
  The amount of energy intake during intervention, conducted with three-day food intake record
Gender and age as independent factor | initial/before intervention
  Subjects gender and age
Personal history as independent factor | initial/before intervention
  Subjects' history that revealed the length of time of diagnosis, and history of previous regular exercise

CONTACTS AND LOCATIONS:
Overall Officials: Nani C Sudarsono, MD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- Center for Sports and Exercise Studies, Indonesian Medical and Research Institute, Faculty of Medicine Universitas Indonesia, Jakarta, Jakarta Pusat, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
IPD is planned to be shared after the completion of study analysis and publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available starting 6 months after publication
Access Criteria: Academics will be able to access information regarding unnamed subject characteristics and intervention detail by sending request to principal investigator. A clearly stated purpose of access will be reviewed.

REFERENCES:
- [Background] Sparks LM, Johannsen NM, Church TS, Earnest CP, Moonen-Kornips E, Moro C, Hesselink MK, Smith SR, Schrauwen P. Nine months of combined training improves ex vivo skeletal muscle metabolism in individuals with type 2 diabetes. J Clin Endocrinol Metab. 2013 Apr;98(4):1694-702. doi: 10.1210/jc.2012-3874. Epub 2013 Mar 5. PMID 23463651
- [Result] Hollekim-Strand SM, Bjorgaas MR, Albrektsen G, Tjonna AE, Wisloff U, Ingul CB. High-intensity interval exercise effectively improves cardiac function in patients with type 2 diabetes mellitus and diastolic dysfunction: a randomized controlled trial. J Am Coll Cardiol. 2014 Oct 21;64(16):1758-60. doi: 10.1016/j.jacc.2014.07.971. No abstract available. PMID 25323267
- [Result] Mitranun W, Deerochanawong C, Tanaka H, Suksom D. Continuous vs interval training on glycemic control and macro- and microvascular reactivity in type 2 diabetic patients. Scand J Med Sci Sports. 2014 Apr;24(2):e69-76. doi: 10.1111/sms.12112. Epub 2013 Sep 17. PMID 24102912
- [Result] Aylin K, Arzu D, Sabri S, Handan TE, Ridvan A. The effect of combined resistance and home-based walking exercise in type 2 diabetes patients. Int J Diabetes Dev Ctries. 2009 Oct;29(4):159-65. doi: 10.4103/0973-3930.57347. PMID 20336198

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-24): https://cdn.clinicaltrials.gov/large-docs/56/NCT03563456/Prot_SAP_000.pdf